CLINICAL TRIAL: NCT06206369
Title: Developing Trustworthy Artificial Intelligence (AI)-Driven Tools to Predict Vascular Disease Risk and Progression
Acronym: VASCULAIDRETRO
Status: Recruiting | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Technical University of Twente (Other); Universidade do Porto (Other); Centre Hospitalier Universitaire de Nice (Other); Stichting Allai (Unknown); University of Belgrade (Other); Brightfish Be (Unknown); Hospital District of Helsinki and Uusimaa (Other); University of Bergen (Other); Asklepios Kliniken Hamburg GmbH (Other); University of Oxford (Other); VINČA INSTITUTE OF NUCLEAR SCIENCES Belgrado (Unknown)
Responsible Party: Principal Investigator, Kak Khee Yeung, M.D., Ph.D., FEBVS, Amsterdam UMC, location VUmc
Other Study IDs: 2011279
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Aneurysm Abdominal; Peripheral Arterial Disease
Keywords: Artificial Intelligence, Prediction models, Image analysis, Abdominal Aortic Aneurysms, Peripheral Arterial Disease
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Peripheral Arterial Disease | interventions — Retrospective Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood and tissue samples (from existing biobanks)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Abdominal Aortic Aneurysm patients
  Interventions: Other: No intervention, retrospective study
- Peripheral Arterial Disease patients
  Interventions: Other: No intervention, retrospective study

INTERVENTIONS:
Other: No intervention, retrospective study — No intervention, retrospective study

SUMMARY:
The VASCULAID-RETRO study, within the broader VASCULAID project, aims to create artificial intelligence (AI) algorithms that can predict cardiovascular events and the progression of abdominal aortic aneurysm (AAA) and peripheral arterial disease (PAD). The study plans to gather and analyze data from at least 5000 AAA and 6000 PAD patients, combining existing cohorts and retrospectively collected data. During this project, AI tools will be developed to perform automatic anatomical segmentation and analyses on multimodal imaging. AI prediction algorithms will be developed based on multisource data (imaging, medical history, -omics).

DETAILED DESCRIPTION:
To date, it is unknown which abdominal aortic aneurysm (AAA) and peripheral arterial disease (PAD) patients will suffer cardiovascular events or in which patients the AAA or PAD will progress. In the VASCULAID project, the VASCULAID-RETRO study aims to leverage data from existing cohorts and retrospectively collected data to develop artificial intelligence (AI) algorithms able to evaluate the risk of cardiovascular events and extent of disease progression.

In order to build and train the algorithms for the predictions, we plan to retrospectively enroll at least 5000 AAA and 6000 PAD patients AI-tools will be applied to the patient data. Automatic anatomical segmentation on images and image analysis on US, CTA and MRI will be performed. Also, algorithms to predict cardiovascular events and AAA or PAD progression based on multi-source data analysis will be developed.

Patient data from European clinical consortium partners is available. This consortium has access to big cohorts with relevant data for the envisioned study that will be used to enrich the existing registries. These data will be used to refine the algorithms developed for the prediction of cardiovascular events and AAA/PAD progression.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 40-90 years old, with an AAA >3cm. This includes patients with infrarenal, juxtarenal, suprarenal, iliac (defined as 1.5x its normal diameter) aneurysms, as well as mycotic aneurysms. Patients that have had interventions or ruptures will also be included
* Males and females, 40-90 years old, all PAD patients (Fontaine stages 1,2,3, and 4).

Exclusion Criteria:

* Patients with an ascending, thoracic, thoracoabdominal (type 1-3) aneurysm.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females between 40 and 90 years of age with an abdominal aortic aneurysm and/or peripheral arterial disease.
Sampling Method: Non-Probability Sample
Enrollment: 11000 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2029-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
Development of disease progression prediction algorithms | 3 years
  The primary goal of this retrospective study is to develop and train algorithms to predict disease progression and risk of cardiovascular events in AAA and PAD patients by leveraging multi-parametric data from 5000 AAA (>1000 in AUMC) and 6000 PAD (>1000 in AUMC) patients from existing cohorts and biobanks.

SECONDARY OUTCOMES:
Internal validation of disease progression prediction algorithms | 3 years
  The secondary objective will be the internal validation of the developed algorithms using data from retrospective cohorts.

CONTACTS AND LOCATIONS:
Locations (6):
- Hospital District of Helsinki and Uusimaa (HUS), Helsinki, Finland
- Asklepios kliniken hamburg, Hamburg, Germany
- Amsterdam UMC, Amsterdam, Netherlands
- University Hospital Center of São João, Porto, Portugal
- University Clinical Centre of Serbia, Belgrade, Serbia
- Oxford University Hospitals, Oxford, United Kingdom

REFERENCES:
- [Derived] Rijken L, Zwetsloot S, Smorenburg S, Wolterink J, Isgum I, Marquering H, van Duivenvoorde J, Ploem C, Jessen R, Catarinella F, Lee R, Bera K, Buisan J, Zhang P, Dias-Neto M, Raffort J, Lareyre F, Muller C, Koncar I, Tomic I, Zivkovic M, Djuric T, Stankovic A, Venermo M, Tulamo R, Behrendt CA, Smit N, Schijven M, van den Born BJ, Delewi R, Jongkind V, Ayyalasomayajula V, Yeung KK. Developing Trustworthy Artificial Intelligence Models to Predict Vascular Disease Progression: the VASCUL-AID-RETRO Study Protocol. J Endovasc Ther. 2025 Feb 7:15266028251313963. doi: 10.1177/15266028251313963. Online ahead of print. PMID 39921236